CLINICAL TRIAL: NCT02091882
Title: OSMITTER 316-13-206A Substudy: A Substudy to Measure the Accuracy of Ingestible Event Marker (IEM) Detection by the Medical Information Device #1 (MIND1) System and Determine the Latency Period
Brief Title: Substudy of the Accuracy of Ingestible Event Marker (IEM) Detection by the Medical Information Device #1 (MIND1)
Acronym: OSMITTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 316-13-206A
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Device Latency
Keywords: OPC-14597 Digital; Aripiprazole; Medical Information Device #1 System (MIND1); Ingestible Event Marker

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Aripiprazole IEM Tablet + Placebo IEM Tablet + MIND1 System (Experimental): Participants were placed a patch by the clinical staff prior to each ingestible event marker (IEM) tablet ingestion. Participants received one IEM tablet approximately every 2 hours, for a total of 4 ingestions on Day 1 at 0, 2, 4 and 6 hours.
  Following placement of the patch by clinic staff, participants ingested one 10 mg aripiprazole-embedded IEM tablet without food at Hour 0, one placebo-embedded IEM tablet without food at approximately Hour 2, one placebo-embedded IEM tablet with a high fat meal at approximately Hour 4, and one placebo-embedded IEM tablet without food at approximately Hour 6. Clinic staff recorded the time of each ingestion of an IEM and the time detected by MIND1 System.
  Interventions: Drug: Placebo; Combination Product: Combination product of Aripiprazole + IEM + Sensor + MIND1 Application

INTERVENTIONS:
Drug: Placebo — Oral placebo-embedded IEM tablet.
Combination Product: Combination product of Aripiprazole + IEM + Sensor + MIND1 Application — Combination product of aripiprazole tablet embedded with sensor and wearable patch with MIND1 system on smartphone
  Other Names: Abilify MyCite®

SUMMARY:
The purpose of this study was to determine the accuracy of IEM detection by the MIND1 System by completing a series of Patch applications and IEM ingestions in the clinic.

DETAILED DESCRIPTION:
The OSMITTER study protocol was designed as a master protocol governing multiple substudies for the rapid assessment of candidate subcomponents for the MIND1 System. This substudy was conducted to determine the accuracy of IEM detection by the MIND1 System by completing a series of Patch applications and IEM ingestions in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy non-pregnant females 18 to 65 years of age at the time of informed consent who are willing to either practice abstinence or 2 barrier methods of birth control or 1 barrier method and an oral contraceptive method
* Participants must be in good general health (not suffering from a serious chronic mental or physical disorder that has required or may in the near future require urgent medical care)
* Body mass index between 19 to 32 kg/m^2
* Ability to eat the high-fat meal

Exclusion Criteria:

* Participants with a history of skin sensitivity to adhesive medical tape or metals
* Participants who, in the opinion of the investigator, is acutely psychotic or manic and has symptoms currently requiring hospitalization
* Participants with a history or evidence of a medical condition that would expose him or her to an undue risk of a significant adverse event (AE) or interfere with assessments of safety during the course of the trial
* Participants have received any investigational product within the last 30 days.
* Participants has a current history of drug or alcohol dependence that meets Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria
* Participants has the presence of cognitive impairment
* Participants currently taking antipsychotic medication
* Participants with a terminal illness
* Participants with a history of chronic dermatitis
* Participants with a history of gastrointestinal surgery that could impair absorption
* Female participants who are breastfeeding and/or who have a positive serum pregnancy test result prior to receiving trial medications
* Sexually active women of childbearing potential (WOCBP) who will not commit to using 2 forms of approved birth control methods or who will not remain abstinent during this trial and for 30 days following the last dose of trial medication
* Sexually active males who will not commit to using 2 of the approved birth control methods or who will not remain abstinent for the duration of the trial and for 90 days following the last dose of trial medication
* No permanent physical residence
* After resting for ≥3 minutes, have a sitting systolic blood pressure <100 or ≥150 millimeters of mercury (mmHg) and/or diastolic blood pressure <50 or ≥90 mmHg
* After resting for ≥3 minutes, have a sitting pulse rate <35 or >100 beats per minute
* Participants who, in the opinion of the investigator, should not participate in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03-21 (Actual); Primary Completion 2014-04-18 (Actual); Study Completion 2014-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Otsuka Pharmaceutical Development & Commercialization
Locations (1):
- Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Jan M, Coppin-Renz A, West R, Gallo CL, Cochran JM, Heumen EV, Fahmy M, Reuteman-Fowler JC. Safety Evaluation in Iterative Development of Wearable Patches for Aripiprazole Tablets With Sensor: Pooled Analysis of Clinical Trials. JMIR Form Res. 2023 Dec 12;7:e44768. doi: 10.2196/44768. PMID 38085556
- [Derived] Rohatagi S, Profit D, Hatch A, Zhao C, Docherty JP, Peters-Strickland TS. Optimization of a Digital Medicine System in Psychiatry. J Clin Psychiatry. 2016 Sep;77(9):e1101-e1107. doi: 10.4088/JCP.16m10693. PMID 27487251
- [Derived] Profit D, Rohatagi S, Zhao C, Hatch A, Docherty JP, Peters-Strickland TS. Developing a Digital Medicine System in Psychiatry: Ingestion Detection Rate and Latency Period. J Clin Psychiatry. 2016 Sep;77(9):e1095-e1100. doi: 10.4088/JCP.16m10643. PMID 27379966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted on 30 healthy participants at one trial site in the United States from 21 March 2014 to 18 April 2014.
Groups:
- Aripiprazole IEM Tablet + Placebo IEM Tablet + MIND1 System: Participants were placed a patch by the clinical staff prior to each ingestible event marker (IEM) tablet ingestion. Participants received one IEM tablet approximately every 2 hours, for a total of 4 ingestions on Day 1 at 0, 2, 4 and 6 hours.
  Following placement of the patch by clinic staff, participants ingested one 10 mg aripiprazole-embedded IEM tablet without food at Hour 0, one placebo-embedded IEM tablet without food at approximately Hour 2, one placebo-embedded IEM tablet with a high fat meal at approximately Hour 4, and one placebo-embedded IEM tablet without food at approximately Hour 6. Clinic staff recorded the time of each ingestion of an IEM and the time it was detected by MIND1 System.
Period: Overall Study
Arm/Group | Aripiprazole IEM Tablet + Placebo IEM Tablet + MIND1 System
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Sample included all participants who ingested at least one aripiprazole + IEM tablet or placebo + IEM tablet.
Groups:
- Aripiprazole IEM Tablet + Placebo IEM Tablet + MIND1 System: Participants were placed a patch by the clinical staff prior to each IEM tablet ingestion. Participants received one IEM tablet approximately every 2 hours, for a total of 4 ingestions on Day 1 at 0, 2, 4 and 6 hours.
  Following placement of the patch by clinic staff, participants ingested one 10 mg aripiprazole-embedded IEM tablet without food at Hour 0, one placebo-embedded IEM tablet without food at approximately Hour 2, one placebo-embedded IEM tablet with a high fat meal at approximately Hour 4, and one placebo-embedded IEM tablet without food at approximately Hour 6. Clinic staff recorded the time of each ingestion of an IEM and the time it was detected by MIND1 System.
Arm/Group | Aripiprazole IEM Tablet + Placebo IEM Tablet + MIND1 System
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Accuracy of Ingestible Event Marker (IEM) Detection
Description: The accuracy of IEM signal detection was collected by comparing the time of ingestion recorded by MIND1 system at different timepoints with the time recorded by the clinic staff. The percentage of participants with the accurate time of IEM detection are reported for each ingestion separately at Hours 0, 2, 4 and 6 on Day 1.
Time Frame: Up to Hour 6 on Day 1
Population: Intention-to-Treat (ITT) Sample included all participants who ingested at least one aripiprazole + IEM tablet, regardless of whether or not ingestion was detected.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Aripiprazole IEM Tablet + Placebo IEM Tablet + MIND1 System
Number analyzed (Participants) | 30
percentage of participants
  Day 1, Hour 0 | 73.3 [57.0 to 86.0]
  Day 1, Hour 2 | 63.3 [46.7 to 77.9]
  Day 1, Hour 4 | 76.7 [60.6 to 88.5]
  Day 1, Hour 6 | 93.3 [80.5 to 98.8]

2. Secondary Outcome: Latency Period From Ingestion to Detection of IEM
Description: Latency period was defined as the time in minutes from the IEM ingestion for both aripiprazole and placebo to the time of detection of IEM by MIND1 system on a smartphone. The latency period is calculated as the difference in the time recorded by the clinic staff of IEM ingestion and the time displayed on the MIND1 application.
Time Frame: Day 1 at Hours 0, 2, 4, 6
Population: ITT Sample included all participants who ingested at least one aripiprazole + IEM tablet, regardless of whether or not ingestion was detected. Number analyzed is the number of participants with data available at specified time points.
Measure: Median (Full Range); unit: minutes
Arm/Group | Aripiprazole IEM Tablet + Placebo IEM Tablet + MIND1 System
Number analyzed (Participants) | 30
minutes
  Day 1, Hour 0: number analyzed (Participants) | 22
  Day 1, Hour 0 | 4 [1 to 14]
  Day 1, Hour 2: number analyzed (Participants) | 19
  Day 1, Hour 2 | 1 [0 to 3]
  Day 1, Hour 4: number analyzed (Participants) | 23
  Day 1, Hour 4 | 1 [0 to 2]
  Day 1, Hour 6: number analyzed (Participants) | 28
  Day 1, Hour 6 | 1 [0 to 4]

ADVERSE EVENTS:
Time Frame: From Day 1 to 2-week safety follow up (Day 15)
Description: Safety Sample included all participants who ingested at least one aripiprazole + IEM tablet or IEM tablet or placebo + IEM tablet.
Arm/Group | Aripiprazole IEM Tablet + Placebo IEM Tablet + MIND1 System
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 5/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole IEM Tablet + Placebo IEM Tablet + MIND1 System (N=30)
Nausea (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.